CLINICAL TRIAL: NCT05860790
Title: Prospective Validation of Clinical Prediction Model for Venous Thromboembolism Following Neurosurgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Zhang, Vice President of Sanbo Brain Hospital, Capital Medical University, Capital Medical University
Other Study IDs: Val. VTE pred. model post-op
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Venous Thromboembolism; Neurosurgery; Risk Assessment
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen refers to biological specimens obtained from patients, such as blood, for routine laboratory tests and analyses, including measurement of coagulation indices, before and after surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Clinical Prediction Model for Venous Thromboembolism Following Neurosurgery — This is a clinical prediction model that uses perioperative clinical indicators and laboratory tests to predict the occurrence of VTE after neurosurgery.

SUMMARY:
Validation of Clinical Prediction Model for Venous Thromboembolism Following Neurosurgery: A Multicenter, Prospective, and Cohort Study

DETAILED DESCRIPTION:
A clinical prediction model for VTE after neurosurgical procedures during hospitalization has been developed and internally retrospectively validated. A multicenter, prospective cohort study is planned to validate this clinical prediction model again.

ELIGIBILITY:
Inclusion Criteria:

1. age >18 years
2. underwent neurosurgical procedures during hospitalization
3. underwent preoperative ultrasound examination

Exclusion Criteria:

1. a patient with obvious bacterial or viral infection within the past two weeks before admission
2. a patient with venous thromboembolism within the past three months before surgery
3. a patient with anticoagulant therapy (direct oral anticoagulants, low molecular weight heparin) was administered continuously or intermittently before admission
4. a patient with a prior coagulation dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients who have undergone neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Symptomatic or asymptomatic VTE | 2023.3-2023.7
  A combination of symptomatic or asymptomatic DVT and symptomatic or asymptomatic PE

SECONDARY OUTCOMES:
DVT | 2023.3-2023.7
  A blood clot within a deep vein, typically in the thigh or leg, which is detected with compressible ultrasound, venography, impedence plethysmography, radiofibrinogen uptake scanning or autopsy based on the time of study. This outcome combines proximal or distal DVT of the leg, upper limb DVT
PE | 2023.3-2023.7
  Obstruction of a pulmonary artery or one of its branches that is usually produced by a blood clot which has originated in a vein of the leg or pelvis and traveled to the lungs, which is diagnosed by CT pulmonary angiography, ventilation-perfusion lung scanning pulmonary angiogram, or by autopsy or equivalent technology based on the time of study. This outcome combines saddle, lobar, segmental or subsegmental PE according to the anatomic location
Proximal DVT | 2023.3-2023.7
  Proximal DVT is a blood clot that is located in the popliteal, femoral, or iliac veins, which is detected with compressible ultrasound, venography, impedence plethysmography, radiofibrinogen uptake scanning or autopsy based on the time of study

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhang, Prof., Principal Investigator — Capital Medical University
Locations (1):
- Sanbo Brain Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided